CLINICAL TRIAL: NCT01415739
Title: Evaluation of a Novel Molecular NSCLC Classification System
Brief Title: Study of Proteins in Tumor Samples From Patients With Non-Small Cell Lung Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Trial closure due to NCI NCTN transition
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-151102; CDR0000706383 (Registry Identifier: NCI Physician Data Query); NCI-2011-02977 (Registry Identifier: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Lung Cancer
Keywords: stage IA non-small cell lung cancer; stage IB non-small cell lung cancer; adenocarcinoma of the lung; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Novel Molecular NSCLC Classification (H & E staining, IHC): Previously collected tissue samples are analyzed via H&E staining and IHC.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research studies protein in tumor samples from patients with non-small cell lung cancer. Finding specific proteins in tumor tissue samples from patients with cancer may help doctors tell what type of lung cancer a patient has and plan better treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To validate a novel 4-protein signature's ability to subtype non-small cell lung cancer (NSCLC) in a treatment-naive, multi-institutional cohort, Cancer and Leukemia Group B (CALGB) 9761.

SECONDARY OBJECTIVES:

I. To estimate the NSCLC misclassification rate in a multi-institutional clinical-trial setting for stage 1 NSCLC (adenocarcinoma versus squamous cell).

OUTLINE:

Previously collected tissue samples are analyzed via hematoxylin and eosin (H&E) staining and immunohistochemistry (IHC).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been registered on CALGB-9761

  * Stage I disease
  * Treatment-naive patients
* A representative paraffin block of the primary tumor must be available from patients on CALGB-9761 and submitted to the CALGB Pathology Coordinating Office
* A separate consent form is not required for this study, as permission for research to be performed on the tissue blocks is included in the consent form for CALGB 9761
* Institutional review board (IRB) review and approval at the institution where the laboratory work will be performed is required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer registered on CALGB 9761
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Validation of a novel 4-protein signature's ability to subtype NSCLC | 1 month

SECONDARY OUTCOMES:
NSCLC misclassification rate | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Boffa, MD, Study Chair — Smilow Cancer Hospital at Yale-New Haven
Locations (1):
- Alliance for Clinical Trials in Oncology, Boston, Massachusetts, United States